CLINICAL TRIAL: NCT06246045
Title: The Impact of System Wide Pulmonary Embolism Screening Program on PERT Activation, Utilization of Advanced Therapies, and 90-Day Outcomes
Brief Title: Artificial Intelligence to StrategiCally Enhance Pulmonary Embolism Response Team Activation
Acronym: ASCENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Closed
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220475
Record Dates: First submitted 2022-02-16; First posted 2024-02-07 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Embolism Subacute Massive
Keywords: PERT; Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early-Invasive Strategy (Experimental): Patients who do not clearly qualify for early intervention (including catheter-directed therapies, systemic thrombolysis, or invasive hemodynamic support) based on assessment by PERT members, will undergo walk testing on the first day of admission. If the subject meets criteria based on pre-specified hemodynamic changes, then the patient will be randomized in a 2:1 fashion to early invasive strategy with catheter-directed therapies as treatment arm.
  Interventions: Diagnostic Test: Walking test
- Traditional Medical Therapy (Active Comparator): Patients who do not clearly qualify for early intervention (including catheter-directed therapies, systemic thrombolysis, or invasive hemodynamic support) based on assessment by PERT members, will undergo walk testing on the first day of admission. If the subject meets criteria based on pre-specified hemodynamic changes, then the patient will be randomized (2:1, treatment to control) to traditional routine care with medical therapy.
  Interventions: Diagnostic Test: Walking test

INTERVENTIONS:
Diagnostic Test: Walking test — PERT will be activated by AI algorithm. As a result of the discussion, patients will either be determined to be appropriate for immediate invasive strategy versus watchful waiting depending on whether high-risk PE criteria are met.
  For those in the intermediate-high risk category, there remains ambiguity on timing and appropriateness of invasive intervention. On day 1 of admission, patients will undergo a walking test evaluating for abnormalities in heart rate, heart rate recovery, and oxygen need. If criteria is met, patients will be randomized in a 2:1 fashion (treatment versus control) to evaluate use of early-invasive strategy.

SUMMARY:
Pulmonary embolism (PE) remains a high mortality and morbidity disease state. The investigators have previously shown that use of a Pulmonary Embolism Response Team (PERT) can improve overall readmission, bleeding, and mortality outcomes. Unfortunately, PERT may still be underutilized from a national standpoint and may not be readily available in underserved areas.

The use of artificial intelligence (AI) may help streamline and systematically ensure unbiased mechanism for activation of PERT for discussion of patients with siginficant clot burden and hemodynamic abnormalities. AI algorithms have been FDA approved for use of triage of the PE patient. The institutional PERT program will adapt the use of an AI algorithm for activation as routine care; the efficiency of activation will be compared to our retrospective historical comparison for efficiency and appropriateness of activation.

The active phase of the study is designed to further differentiate between patients who are considered to be intermediate-high risk category but yet do not clearly qualify for invasive therapy (catheter-directed therapy, systemic thrombolysis, or invasive hemodynamic support). These patients will undergo walking test to further understand noninvasive hemodynamic compromise and undergo 2:1 randomization to early-invasive strategy versus mtranditional medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients obtaining a CT at University Hospitals found to have a pulmonary embolism with evidence of right ventricular strain (RV:LV > 0.9) along with an abnormal vital sign (HR > 110 bpm, RR > 30/min, SBP < 100 mmHg, or O2 saturation < 90%)
* Patients undergoing PERT discussion as deemed appropriate by the provider

Exclusion Criteria:

* Age <18
* Pregnant patients. Women of childbearing age will be asked if they are pregnant before enrollment. No formal pregnancy test will be performed as a part of this study. If a patient does require invasive intervention, as part of the routine procedure for cardiac catheterization laboratory, women of childbearing age will either undergo pregnancy testing or opt-out per their own discretion
* Patients unable to perform 6MWT (e.g., lack of one or both legs) will not be included in the randomization. They will be included in the observation for routine treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-activation | 3 days
  Activation of PERT from time of CT scan to call; compared to historical control

SECONDARY OUTCOMES:
Length of stay | 30 days
  Total length of hospital stay
6-minute walk test (6MWT) | 6 minutes
  The distance (meter) and walking speed (meter per seconds) in a 6-minute walk test.
Change in quality of life as measured by PEmb QoL | Baseline, 30 days, 90 days
  PEmb-QoL summary score (0-100, higher score indicate worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacey MJ, Hammad TA, Parikh M, Tefera L, Sharma P, Kahl R, Zemko A, Li J, Carman T, Schilz R, Shishehbor MH. Prospective Experience of Pulmonary Embolism Management and Outcomes. J Invasive Cardiol. 2021 Mar;33(3):E173-E180. Epub 2021 Feb 11. PMID 33570502
- [Background] Parikh M, Chahine NM, Hammad TA, Tefera L, Li J, Carman T, Schilz R, Shishehbor MH. Predictors and potential advantages of PERT and advanced therapy use in acute pulmonary embolism. Catheter Cardiovasc Interv. 2021 Jun 1;97(7):1430-1437. doi: 10.1002/ccd.29697. Epub 2021 Apr 12. PMID 33844438